CLINICAL TRIAL: NCT04652960
Title: A Phase I Study With an Expansion Cohort of Duvelisib and Nivolumab in Mycosis Fungoides (MF) and Sézary Syndrome (SS)
Brief Title: Duvelisib and Nivolumab for the Treatment of Stage IIB-IVB Mycosis Fungoides and Sezary Syndrome
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-11641; NCI-2020-11641 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10347 (Other: Yale University Cancer Center LAO); 10347 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2020-12-03; First posted 2020-12-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Stage IIB Mycosis Fungoides and Sezary Syndrome AJCC v8; Stage III Mycosis Fungoides and Sezary Syndrome AJCC v8; Stage IV Mycosis Fungoides and Sezary Syndrome AJCC v8
MeSH Terms: conditions — Mycosis Fungoides; Sezary Syndrome | interventions — Specimen Handling; duvelisib; Nivolumab; Magnetic Resonance Spectroscopy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (duvelisib, nivolumab) (Experimental): Patients receive duvelisib PO QD or BID on days 1-28 or days 1-14 and nivolumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo PET-CT or CT scan at baseline. Patients also undergo punch biopsy and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Duvelisib; Biological: Nivolumab; Procedure: Positron Emission Tomography; Procedure: Punch Biopsy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Duvelisib — Given PO
  Other Names: 8-Chloro-2-phenyl-3-((1S)-1-(7H-purin-6-ylamino)ethyl)isoquinolin-1(2H)-one; Copiktra; INK-1197; IPI 145; IPI-145; IPI145
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: Punch Biopsy — Undergo punch biopsies
  Other Names: BIOPSY, PUNCH; Punch Biopsy of Skin

SUMMARY:
This phase I trial identifies the best dose, possible benefits, and/or side effects of duvelisib in combination with nivolumab in treating patients with stage IIB-IVB mycosis fungoides and Sezary syndrome. Duvelisib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving duvelisib in combination with nivolumab may work better than giving each of these drugs individually, or treating with the usual approach in patients with mycosis fungoides and Sezary syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the recommended phase II dose (RP2D) or maximum tolerated dose (MTD) of the combination of duvelisib with nivolumab in patients with advanced mycosis fungoides/Sezary syndrome (MF/SS).

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. Ia. To determine the overall response rate at four months to the combination of nivolumab and duvelisib.

Ib. To determine the time to maximum response, best overall response rate, complete remission rate, and duration of response among responding patients.

EXPLORATORY OBJECTIVES:

I. To evaluate whether intra-patient changes in serum cytokines (soluble CD40L, TNF-beta, IL-17alpha, IL-15, CXCL13, IL-12p40) predict response to duvelisib in combination with nivolumab in cutaneous T-cell lymphoma (CTCL).

II. To explore whether the combination of duvelisib and nivolumab changes the T-cell repertoire including T-cell receptor sequencing pre- and post- treatment with duvelisib and nivolumab in effort to better understand skin flare and other immunogenic reactions to this combination therapy.

OUTLINE: This is a dose-escalation study of duvelisib in combination with fixed dose nivolumab followed by a dose-expansion study.

Patients receive duvelisib orally (PO) once daily (QD) or twice daily (BID) on days 1-28 or days 1-14 and nivolumab intravenously (IV) over 30 minutes on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo positron emission tomography (PET)-computed tomography (CT) or CT scan at baseline. Patients also undergo punch biopsy and collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed MF or SS, stages IIB to IVB with measurable disease and/or detectable blood involvement based on the Global Cutaneous Lymphoma Response Criteria
* Patients must have had at least one line of prior systemic therapy
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of duvelisib in combination with nivolumab in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 50%)
* Absolute neutrophil count >= 1000/mcL
* Platelets > 75,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) or =< 5 x institutional ULN if with history of Gilbert's syndrome
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
* Creatinine =< 2.0 x institutional ULN
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* The effects of nivolumab and duvelisib on the developing human fetus are unknown. For this reason and because other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. WOCBP should use an adequate method to avoid pregnancy for 5 months after the last dose of nivolumab and duvelisib. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 7 days prior to the start of nivolumab and duvelisib. Women must not be breastfeeding. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and duvelisib and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational product. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile as well as azoospermic men) do not require contraception. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL
* Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 7 months after completion of administration of investigational agents on this study
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial

Exclusion Criteria:

* Prior therapy with a PI3K inhibitor
* Prior therapy with nivolumab or other agents targeting T-cell co-stimulation or checkpoint pathways
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded. These include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease. Patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible. Patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible
* Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event)
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 7 days of study drug administration. Inhaled or topical steroids, steroids for physiologic or adrenal replacement doses =< 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* History of tuberculosis treatment within the 2 years prior to enrollment
* Ongoing treatment with other immunosuppressive agent including, but not limited to, methotrexate, azathioprine, anti-tumor necrosis factor (TNF) agents, etc. with the exception of steroids
* Administration of a live or live attenuated vaccine within 6 weeks of initiation of study therapy
* Ongoing treatment with systemic steroids at dose equivalent to greater than prednisone 10 mg daily or other immunosuppressive medication within 7 days of initiation of study therapy

  * Inhaled steroids will be permitted
  * Topical steroids for cutaneous manifestations of MF/SS will be permitted below:

    * Continued use of select concomitant topical steroids is permitted if the patient has remained clinically stable for at least 4 weeks.
    * Patients who are on low or moderate potency topical corticosteroids may participate if they are on a stable dose for at least 4 weeks before enrollment. Local injections of corticosteroids are acceptable; all corticosteroids will be reported as concomitant medications.
  * Patients prescribed prednisone 10 mg PO daily or less (or equivalent) will not be excluded
* Concomitant use of another systemic therapy for MF/SS. Patients must have the following minimum wash-out from previous treatments:

  * At least 8 weeks for low-dose (12 Gy or less) total skin electron beam therapy (TSEBT)
  * At least 4 weeks for systemic cytotoxic anticancer agents or for tumor-targeting monoclonal antibodies (mAbs), with the exception of alemtuzumab, for which the washout is at least 16 weeks
  * At least 2 weeks or 5 half-lives for systemic retinoids, interferons, vorinostat, romidepsin, and denileukin diftitox, or anticancer investigational agents that are not defined as immunotherapy
  * At least 2 weeks for local radiation therapy
  * At least 1 week for topical retinoids, nitrogen mustard, or imiquimod
* Concomitant malignancy requiring active systemic therapy, excluding adjuvant endocrine therapy with the following exceptions:

  * Patients with non-melanoma skin cancer or carcinoma in situ of the cervix will not be excluded
  * Adjuvant or maintenance therapy to reduce the risk of recurrence of another malignancy (excluding cutaneous T-cell lymphoma) is permissible after discussion with the Washington University principal investigator
  * Subjects with previous malignancies are eligible if disease-free for > 2 years
* History of solid organ transplantation or allogeneic bone marrow transplantation
* Uncontrolled infection requiring systemic antimicrobials: Patients on antibacterial, antifungal, and antiviral prophylaxis will not be excluded if all other exclusion / inclusion criteria are met
* Patients with active cytomegalovirus (CMV) (positive serology for anti-CMV IgM antibody and negative for anti-CMV IgG antibody or positive CMV PCR with clinical manifestations consistent with active CMV infection) and requiring therapy will be excluded from participation in the study. Carriers will be monitored per institutional guidelines
* Patients should be excluded if they have known active hepatitis B (e.g. hepatitis B virus [HBV] surface antigen [HBsAg] reactive) or hepatitis C (e.g. hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)

  * Patients with chronic HBV or HCV are defined as patients with positive hepatitis B serology: Patients with a negative HBsAg and a positive hepatitis B core antibody (HBcAb) require an undetectable/negative hepatitis B deoxyribonucleic acid (DNA) test (e.g. polymerase chain reaction [PCR] test) to be enrolled, and will require prophylactic antiviral treatment initiated prior to the first dose of study drug, and continued until approximately 6 to 12 months after completion of study drug(s)
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1), with the exception of alopecia and neuropathy
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to duvelisib or nivolumab
* Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 are ineligible to start study therapy. Patients who are on strong inhibitors or inducers of CYP3A4 may start study therapy if discontinued 5 half lives before start of study therapy. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, interstitial lung disease or active, non-infectious pneumonitis, congestive heart failure New York Heart Association (NYHA) grade >= 3, unstable angina pectoris, and cardiac arrhythmia
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Baseline QT interval corrected with Fridericia's method (QTcF) > 500 ms

  * Note: Criteria does not apply to subjects with a right or left bundle branch block
* Pregnant women are excluded from this study because nivolumab and duvelisib have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with nivolumab and duvelisib, breastfeeding should be discontinued if the mother is treated with nivolumab and duvelisib. These potential risks may also apply to other agents used in this study
* Patients who have had evidence of active or acute diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation should be evaluated for the potential need for additional treatment before coming on study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2026-12-03 (Estimated); Study Completion 2026-12-03 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose or recommended phase II dose (RP2D) | Through completion of 3 cycles (each cycle is 28 days)
  If one dose-limiting toxicity (DLT) is seen in the first three patients treated at a given dose level, then three additional patients will be evaluated at that same dose level. If DLTs are present at < 2 of 6 patients, the next dose level will be explored. If 3 patients are treated at the maximal dose level without DLT, three more patients will be enrolled to that dose level to evaluate for DLT. If < 2/6 DLTs are seen at that dose level, it will be deemed the RP2D.
Incidence of adverse events | For 30 days after last dose of study treatment or until the initiation of alternative treatment, whichever comes first. If removed for an adverse event, the adverse event causing removal will be followed until resolution or stabilization

SECONDARY OUTCOMES:
Overall response rate (ORR) | At 4 months
  Defined as the proportion of patients having achieved partial response (PR) or complete response (CR) at any time prior to the four-month time point. ORR will be estimated as a sample proportion with a 95% confidence interval using the method of Agresti and Coull around the point estimate. Will be assessed using the Global Response Criteria for cutaneous T-cell lymphoma which includes a skin-based assessment (modified severity-weighted assessment tool), peripheral blood evaluation for circulating Sezary cells by flow cytometry, and radiographic evaluation (contrast-enhanced computed tomography [CT] chest/abdomen/pelvis or positron emission tomography [PET]/CT).
Complete response rate (CRR) | Up to 2 years post-treatment
  Defined as the percentage of patients who achieve CR at any timepoint. CRR will be estimated as a sample proportion with associated confidence intervals.
Overall response rate (ORR) for all treated patients | Up to 2 years post-treatment
  Defined as the percentage of patients who achieve CR or PR at any timepoint. ORR will be estimated as a sample proportion with associated confidence intervals. Will be assessed using the Global Response Criteria for cutaneous T-cell lymphoma which includes a skin-based assessment (modified severity-weighted assessment tool), peripheral blood evaluation for circulating Sezary cells by flow cytometry, and radiographic evaluation (contrast-enhanced CT chest/abdomen/pelvis or PET/CT).
Disease control rate (DCR) | At 4 months
  Defined as the proportion of patients who achieve CR, PR, or stable disease (SD) at the four-month time point. DCR will be estimated as a sample proportion with associated confidence intervals.
Duration of response (DOR) for responding patients | From the first documentation of response to the first documentation of progressive disease (PD) or death due to any cause, assessed up to 2 years post-treatment
  DOR will be determined on intention-to-treat basis and will be estimated using Kaplan-Meier analysis.
Time to maximum response among responding patients | From study enrollment to time of documentation of either PR (if PR is the best response achieved) or CR (if CR is the best response achieved), assessed up to 2 years post-treatment
  Time to maximum response will be determined on intention-to-treat basis and will be estimated using Kaplan-Meier analysis.
Overall survival (OS) | From study enrollment to death from any cause, assessed up to 2 years post-treatment
  OS will be determined on intention-to-treat basis and will be estimated using Kaplan-Meier analysis.
Progression-free survival (PFS) | From study enrollment to first documentation of PD, assessed up to 2 years post-treatment
  PFS will be determined on intention-to-treat basis and will be estimated using Kaplan-Meier analysis.

OTHER OUTCOMES:
Change in the immune composition | Before the start of treatment, on treatment, at end of treatment, and at the time of flare, up to 2 years post-treatment
  Will evaluate the changes in the immune composition by CyTOF and MIBI and in serum cytokine profiles (Olink) on samples before the start of treatment, on treatment, at end of treatment, and at the time of flare. For comparing biomarkers pre- and post-treatment we will use paired Wilcoxon signed-rank tests for each marker comparing to baseline earlier timepoints. Will correct for multiple hypothesis testing using the Benjamini-Hochberg procedure. Will also use logistic regression to assess the relationship between biomarkers and response.

CONTACTS AND LOCATIONS:
Overall Officials: Neha Mehta-Shah, Principal Investigator — Yale University Cancer Center LAO
Locations (17):
- United States (17):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2025-07-29): https://cdn.clinicaltrials.gov/large-docs/60/NCT04652960/ICF_000.pdf